CLINICAL TRIAL: NCT06360341
Title: Feasibility and Acceptability of an Emergency Department Digital Pain Self-Management Intervention to Improve Acute Low Back Pain Outcomes: A Pilot Randomized Controlled Trial
Brief Title: Emergency Department Digital Pain Self-Management Intervention to Improve Acute Low Back Pain Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202301946
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-11

CONDITIONS: Low Back Pain, Mechanical; Acute Pain
Keywords: Pilot Randomized Controlled Trial; Digital Pain Self-Management Intervention; Improving Health Outcomes
MeSH Terms: conditions — Low Back Pain; Acute Pain

STUDY DESIGN:
Intervention Model Description: Individuals in the pilot randomized controlled trial (RCT) intervention will be randomized to either the intervention or routine discharge care (RC) using REDCap randomizer and assigned to RC or Emergency Department Digital Pain Self-Management Intervention (EDPSI) + RC.
Masking Description: Randomization to RC or Intervention group will not be masked to the Principal Investigator (PI), co-PI, or to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive Emergency Department Digital Pain Self-Management Intervention (EDPSI) + routine discharge care (RC).
  Interventions: Behavioral: Emergency Department Digital Pain Self-Management Intervention (EDPSI); Other: Routine Discharge Care
- Control Group (Active Comparator): The control group will receive routine discharge care (RC).
  Interventions: Other: Routine Discharge Care

INTERVENTIONS:
Behavioral: Emergency Department Digital Pain Self-Management Intervention (EDPSI) — The EDPSI is a developed supplemental digital video for patients presenting to the emergency department with acute low back pain (aLBP). The content consists of self-management approaches for diverse adult patient preferences including biopsychosocial contributors to pain and clinical practice guidelines to self-management options. Highlights of the discharge instructions summary include follow-up with provider, red flag warnings, and medication safety. Actor demonstration of ergonomics and range of motion movements provide application of Physical Therapy (PT)-based preventative strategies. Combination therapies including PT counseling, complementary alternative medicine (acupuncture, massage, yoga, or Pilates), and use of and safety with ice or heat thermal therapies. Active participation, stress management, and involvement of support systems are addressed.
  Arms: Intervention Group
Other: Routine Discharge Care — Routine Discharge Care

SUMMARY:
The proposed study aims to evaluate a pilot emergency department (ED) digital pain self-management intervention (EDPSI) focused on improving self-efficacy, knowledge, and skills, thus reducing the transition from acute to chronic low back pain in ED patients discharged with axial acute low back pain (aLBP). The proposed research has significant potential to improve self-efficacy (the confidence in one's ability to manage their condition) which is one of the most potent factors for improved health outcomes.

DETAILED DESCRIPTION:
Investigators:

Principal Investigator: Alexandria Carey (University of Florida, PhD Candidate) Co-Investigator/ Supervisory Chair: Ann Horgas

Supervisory Committee Members:

* Laurie Duckworth
* Hwayoung Cho
* Jason M. Beneciuk Previous Co-Investigator (2022-2024): Angela Starkweather

IRB #: 202301946

Study Site: UF Health Emergency Centers, campuses in Gainesville, Florida

Study Sponsor: University of Florida

Background/Significance: Over 3.4 million acute axial low back pain (aLBP) cases are treated annually in the United States (US) emergency departments (ED). ED patients with aLBP receive varying verbal and written discharge routine care (RC), leading to gaps in patient discharge effectiveness and effective self-management. Ineffective aLBP self-management may increase the risk of transition to chronic low back pain (cLPB), a chief cause of worldwide disability, with associated costs reaching > $60 million annually. This research will address this significant problem by evaluating an ED digital pain self-management intervention (EDPSI) focused on improving self-efficacy, knowledge, and skills, thus reducing the transition from aLBP to cLBP in ED patients discharged with axial aLBP. The proposed research has significant potential to increase self-efficacy, which is one of the most potent mechanisms of behavior change and improved health outcomes. Due to the focus on accessibility and usability, the intervention may reduce discharge disparities in aLBP self-management, especially among patients with low health literacy.

Study Questions: This research will answer the following questions: 1) Will an ED digital pain self-management intervention (EDPSI) focused on improving self-efficacy, knowledge retention, and skills progress patient self-management behaviors and health status?

Primary Objective: Primary Aims 1.1.1 Evaluate the feasibility and acceptability of an ED digital pain self-management intervention (EDPSI) for individuals aged 18 years and older presenting to the ED with acute axial low back pain (aLPB).

* Feasibility will be measured by appropriateness, relevance to the ED population, recruitment, retention, and engagement percentages using the following criteria:

  * Of patients who meet eligibility criteria for the study, >80% will voluntarily consent to participate in the study.
  * Of patients consented to the study, >80% will complete the 1-week follow up measures.
  * Of patients randomized to the intervention group, >70% will attend booster sessions at 2 and 8 weeks.
  * Of patients randomized to the intervention group, >80% will recall the discharge video content during booster sessions at 2 and 8 weeks.
* Acceptability of the intervention will be evaluated using the Preference and Satisfaction Questionnaire (EPSQ) and Patient Satisfaction and Healthcare Utilization Questionnaire (PSHU) post-intervention and the following criteria:

  * Of patients who complete the study, >80% will rate the intervention as "satisfactory" or "highly satisfactory"
  * Of patients who complete the study, >80% would be willing to refer a friend or family member with acute low back pain to the intervention.
  * Of overall patients who complete the study, >80% would be satisfied with study participation and be willing to recommend the study.

1.1.2 Evaluate the preliminary clinical efficacy of the EDPSI on participant's self-management, pain self-efficacy, severity, and interference. Self-management, defined as participant engagement in self-management behaviors and integration into lifestyle by acknowledging confidence and demonstrating knowledge retainment and skills in managing to perform everyday activities while in acute pain. Preliminary clinical efficacy would be assessed using estimates of Minimal Clinically Important Difference (MCID), the smallest change in an outcome that patients perceive as meaningful and indicative of improvement.

* Self-management (self-efficacy, knowledge, and skills) preliminary clinical efficacy (MCID) will be measured using the 13-item Patient Activation Measure (PAM) at 1-week, 6-weeks, and 12-weeks.
* Self-efficacy (confidence) preliminary clinical efficacy (MCID) will be measured using the Pain Self-Efficacy Questionnaire (PSEQ) at 1-week, 6-weeks, and 12-weeks.
* Pain severity and interference preliminary clinical efficacy (MCID) will be measured using the Brief Pain Inventory-Short Form (BPI-SF) at 1-week, 6-weeks, and 12-weeks.

Methods: The proposed phased study will use a two-group pilot randomized controlled trial design to enroll 30 individuals who have been seen in the ED with aLBP. Participants will be randomized into RC or RC + EDPSI and receive follow-up surveys for 12-weeks post-intervention. The intervention group will also receive Booster sessions via Zoom with the principal investigator to assess and reinforce their knowledge retention of techniques and provide return demonstration reinforcement ergonomics and range of motion movements demonstrated, in weeks two and eight.

Outcome Measures: All participants will be followed for 12-weeks assessing self-management and self-efficacy in weeks 1, 6, and 12. Feasibility will be measured by recruitment, enrollment, and retention percentages. Acceptability and education satisfaction will be measured using the Education-Preference and Satisfaction Questionnaire (EPSQ) post-intervention. Self-management sustainment will be measured including PSEQ, PAM, and patient satisfaction and healthcare utilization (PSHU) requesting patient overall satisfaction, additional healthcare utilization, and pain management related to continued back pain or complications post-injury.

ELIGIBILITY:
Inclusion Criteria:

* Patient subjective chief complaint of acute or subacute axial low back pain, low back injury, mechanical low back pain, non-specific low back pain, back sprain, or back strain Or
* Provider diagnosis of acute axial low back pain
* ICD-10 discharge codes:
* Low back pain, unspecified M54.50
* Pain of lumbar, acute, for less than 3 months; low back strain (S39.012)
* Unspecific injury of lower back, initial encounter (S39.92XA) And
* Are aged 18 years and older
* Can read and consent to participate in the trial
* Can read and speak English
* Can complete study follow-up at prespecified intervals
* Have access to Wi-Fi
* Have access to a phone or other smart device (e.g. a smartphone, tablet, or computer) that would allow receiving of phone calls, text messages, Zoom meetings, or emails

Exclusion Criteria:

* Admission to the hospital
* Disabilities that would inhibit digital intervention learning (medical, psychiatric, traumatic brain injury, concussion, blindness, or deaf)
* Prisoners/Incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Improving Self-Management Health Outcomes | 12-weeks
  Feasibility and Acceptability of the pilot study will assess recruitment, retention, engagement, satisfaction, and willingness to recommend. Acceptability and intervention satisfaction will be assessed using the Education Preference and Satisfaction Questionnaire (EPSQ) and study satisfaction and recommendation using the Patient Satisfaction and Healthcare Utilization Questionnaire (PSHU). Preliminary Clinical Efficacy will be assessed for self-management, self-efficacy, pain severity and interference. Self-management will be assessed using the short 13-item Patient Activation Measure (PAM), self-efficacy using the Pain Self-Efficacy Questionnaire (PSEQ), pain severity and interference using the Brief Pain Inventory Short-Form (BPI-SF). Preliminary clinical efficacy of the EDPSI for adults with aLBP will be evaluated using estimates of Minimal Clinically Important Difference (MCID), the smallest change in an outcome that patients perceive as meaningful and indicative of improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandria A Carey, MSN, MBA, Principal Investigator — University of Florida
Locations (1):
- UF Health Emergency Centers, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Data Integrity and Oversight: The PI will be responsible for the ethical conduct of the study by all federal, state, and local laws and regulations, institutional policies, and the requirements of the IRB.
  Data Management: Subject confidentiality is strictly held in trust by the investigators and study staff. All written informed consent forms will be immediately secured in the locked and secured office of the PI in a locked and secured study-designated cabinet in the College of Nursing Room 2203. Study data collection and instrument administration will be conducted via REDCap, a secure, web-based application designed to support data capture, providing 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical Packages; and 4) procedures for importing data from external sources. REDCap has built-in measures to protect participants' anonymity.

REFERENCES:
- [Background] Anderson JK, Wallace LM. Evaluation of uptake and effect on patient-reported outcomes of a clinician and patient co-led chronic musculoskeletal pain self-management programme provided by the UK National Health Service. Br J Pain. 2018 May;12(2):104-112. doi: 10.1177/2049463717734015. Epub 2017 Sep 26. PMID 29796262
- [Background] Baker TL, Greiner JV. Guidelines: Discharge Instructions for Covid-19 Patients. J Prim Care Community Health. 2021 Jan-Dec;12:21501327211024400. doi: 10.1177/21501327211024400. PMID 34142617
- [Background] Boden-Albala B, Goldmann E, Parikh NS, Carman H, Roberts ET, Lord AS, Torrico V, Appleton N, Birkemeier J, Parides M, Quarles L. Efficacy of a Discharge Educational Strategy vs Standard Discharge Care on Reduction of Vascular Risk in Patients With Stroke and Transient Ischemic Attack: The DESERVE Randomized Clinical Trial. JAMA Neurol. 2019 Jan 1;76(1):20-27. doi: 10.1001/jamaneurol.2018.2926. PMID 30304326
- [Background] Chidume T, Pass-Ivy S. Student-Novice Nurse Preparation: Addressing Barriers in Discharge Teaching. Nurs Educ Perspect. 2020 Mar/Apr;41(2):88-91. doi: 10.1097/01.NEP.0000000000000498. PMID 31107815
- [Background] DeSai C, Janowiak K, Secheli B, Phelps E, McDonald S, Reed G, Blomkalns A. Empowering patients: simplifying discharge instructions. BMJ Open Qual. 2021 Sep;10(3):e001419. doi: 10.1136/bmjoq-2021-001419. PMID 34521621
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. J Pain. 2014 Jun;15(6):569-85. doi: 10.1016/j.jpain.2014.03.005. Epub 2014 Apr 29. PMID 24787228
- [Background] Dube MO, Langevin P, Roy JS. Measurement properties of the Pain Self-Efficacy Questionnaire in populations with musculoskeletal disorders: a systematic review. Pain Rep. 2021 Dec 21;6(4):e972. doi: 10.1097/PR9.0000000000000972. eCollection 2021 Nov-Dec. PMID 34963996
- [Background] Edwards J, Hayden J, Asbridge M, Magee K. The prevalence of low back pain in the emergency department: a descriptive study set in the Charles V. Keating Emergency and Trauma Centre, Halifax, Nova Scotia, Canada. BMC Musculoskelet Disord. 2018 Aug 23;19(1):306. doi: 10.1186/s12891-018-2237-x. PMID 30134874
- [Background] George SZ, Fritz JM, Silfies SP, Schneider MJ, Beneciuk JM, Lentz TA, Gilliam JR, Hendren S, Norman KS. Interventions for the Management of Acute and Chronic Low Back Pain: Revision 2021. J Orthop Sports Phys Ther. 2021 Nov;51(11):CPG1-CPG60. doi: 10.2519/jospt.2021.0304. PMID 34719942
- [Background] Gilmore AK, Walsh K, Frazier P, Ledray L, Acierno R, Ruggiero KJ, Kilpatrick DG, Resnick HS. Prescription Opioid Misuse After a Recent Sexual Assault: A Randomized Clinical Trial of a Video Intervention. Am J Addict. 2019 Sep;28(5):376-381. doi: 10.1111/ajad.12922. Epub 2019 Jun 26. PMID 31242340
- [Background] Gold JM, Chadwick W, Gustafson M, Valenzuela Riveros LF, Mello A, Nasr A. Parent Perceptions and Experiences Regarding Medication Education at Time of Hospital Discharge for Children With Medical Complexity. Hosp Pediatr. 2020 Aug;10(8):679-686. doi: 10.1542/hpeds.2020-0078. PMID 32737165
- [Background] Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Serv Res. 2005 Dec;40(6 Pt 1):1918-30. doi: 10.1111/j.1475-6773.2005.00438.x. PMID 16336556
- [Background] Hodges R, Stepien S, Kim LY. Quality Improvement: Using Teach-Back to Improve Patient Satisfaction during Discharge in the Emergency Department. J Emerg Nurs. 2021 Nov;47(6):870-878. doi: 10.1016/j.jen.2021.05.006. Epub 2021 Jun 30. PMID 34215436
- [Background] Hoek AE, Geraerds AJLM, Rood PPM, Joosten M, Dippel DWJ, van Beeck EF, van den Hengel L, Dijkstra B, Papathanasiou D, van Rijssel D, van den Hamer M, Schuit SCE, Burdorf A, Haagsma JA, Polinder S. The Effect of Written and Video Discharge Instructions After Mild Traumatic Brain Injury on Healthcare Costs and Productivity Costs. J Head Trauma Rehabil. 2022 Jul-Aug 01;37(4):E231-E241. doi: 10.1097/HTR.0000000000000720. Epub 2021 Jul 26. PMID 34320553
- [Background] In J. Introduction of a pilot study. Korean J Anesthesiol. 2017 Dec;70(6):601-605. doi: 10.4097/kjae.2017.70.6.601. Epub 2017 Nov 14. PMID 29225742
- [Background] Kim HS, Muschong KM, Fishman IL, Schauer JM, Seitz AL, Strickland KJ, Lambert BL, McCarthy DM, Vu MH, Ciolino JD. Embedded emergency department physical therapy versus usual care for acute low back pain: a protocol for the NEED-PT randomised trial. BMJ Open. 2022 May 24;12(5):e061283. doi: 10.1136/bmjopen-2022-061283. PMID 35613820
- [Background] Keenan RP, Lovanio K, Lapidus G, Chenard D, Smith S. Improved Concussion Discharge Instructions in a Pediatric Emergency Department. Adv Emerg Nurs J. 2020 Jan/Mar;42(1):63-70. doi: 10.1097/TME.0000000000000280. PMID 32000192
- [Background] Newnham H, Barker A, Ritchie E, Hitchcock K, Gibbs H, Holton S. Discharge communication practices and healthcare provider and patient preferences, satisfaction and comprehension: A systematic review. Int J Qual Health Care. 2017 Oct 1;29(6):752-768. doi: 10.1093/intqhc/mzx121. PMID 29025093
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Oliveira CB, Hamilton M, Traeger A, Buchbinder R, Richards B, Rogan E, Maher CG, Machado GC. Do Patients with Acute Low Back Pain in Emergency Departments Have More Severe Symptoms than Those in General Practice? ASystematic Review with Meta-Analysis. Pain Med. 2022 Apr 8;23(4):614-624. doi: 10.1093/pm/pnab260. PMID 34480571
- [Background] Pellet J, Weiss M, Zuniga F, Mabire C. Implementation and preliminary testing of a theory-guided nursing discharge teaching intervention for adult inpatients aged 50 and over with multimorbidity: a pragmatic feasibility study protocol. Pilot Feasibility Stud. 2021 Mar 17;7(1):71. doi: 10.1186/s40814-021-00812-4. PMID 33731212
- [Background] Peyman H, Sadeghifar J, Khajavikhan J, Yasemi M, Rasool M, Yaghoubi YM, Nahal MM, Karim H. Using VARK Approach for Assessing Preferred Learning Styles of First Year Medical Sciences Students: A Survey from Iran. J Clin Diagn Res. 2014 Aug;8(8):GC01-4. doi: 10.7860/JCDR/2014/8089.4667. Epub 2014 Aug 20. PMID 25302208
- [Background] Platts-Mills TF, McLean SA, Weinberger M, Stearns SC, Bush M, Teresi BB, Hurka-Richardson K, Kroenke K, Kerns RD, Weaver MA, Keefe FJ. Brief educational video plus telecare to enhance recovery for older emergency department patients with acute musculoskeletal pain: study protocol for the BETTER randomized controlled trial. Trials. 2020 Jul 6;21(1):615. doi: 10.1186/s13063-020-04552-3. PMID 32631400
- [Background] Ryan P, Sawin KJ. The Individual and Family Self-Management Theory: background and perspectives on context, process, and outcomes. Nurs Outlook. 2009 Jul-Aug;57(4):217-225.e6. doi: 10.1016/j.outlook.2008.10.004. PMID 19631064
- [Background] Urits I, Burshtein A, Sharma M, Testa L, Gold PA, Orhurhu V, Viswanath O, Jones MR, Sidransky MA, Spektor B, Kaye AD. Low Back Pain, a Comprehensive Review: Pathophysiology, Diagnosis, and Treatment. Curr Pain Headache Rep. 2019 Mar 11;23(3):23. doi: 10.1007/s11916-019-0757-1. PMID 30854609
- [Background] Vayngortin T, Bachrach L, Patel S, Tebb K. Adolescents' Acceptance of Long-Acting Reversible Contraception After an Educational Intervention in the Emergency Department: A Randomized Controlled Trial. West J Emerg Med. 2020 Apr 21;21(3):640-646. doi: 10.5811/westjem.2020.2.45433. PMID 32421513
- [Background] Wang C, Lang J, Xuan L, Li X, Zhang L. The effect of health literacy and self-management efficacy on the health-related quality of life of hypertensive patients in a western rural area of China: a cross-sectional study. Int J Equity Health. 2017 Jul 1;16(1):58. doi: 10.1186/s12939-017-0551-9. PMID 28666443
- [Background] Waszak DL, Mitchell AM, Ren D, Fennimore LA. A Quality Improvement Project to Improve Education Provided by Nurses to ED Patients Prescribed Opioid Analgesics at Discharge. J Emerg Nurs. 2018 Jul;44(4):336-344. doi: 10.1016/j.jen.2017.09.010. Epub 2017 Oct 27. PMID 29107318
- [Background] Wilkin ZL. Effects of Video Discharge Instructions on Patient Understanding: A Prospective, Randomized Trial. Adv Emerg Nurs J. 2020 Jan/Mar;42(1):71-78. doi: 10.1097/TME.0000000000000279. PMID 32000193
- [Background] Wray A, Goubert R, Gadepally R, Boysen-Osborn M, Wiechmann W, Toohey S. Utilization of Educational Videos to Improve Communication and Discharge Instructions. West J Emerg Med. 2021 Apr 27;22(3):644-647. doi: 10.5811/westjem.2021.1.48968. PMID 34125040
- See also: Pain self-efficacy questionnaire (PSEQ). — https://novopsych.com.au/assessments/health/pain-self-efficacy-questionnaire-pseq/
- See also: FastStats - emergency department visits. Centers for Disease Control and Prevention. — https://www.cdc.gov/nchs/fastats/emergency-department.htm
- See also: Understanding statistical power and significance testing - an interactive visualization. — https://rpsychologist.com/d3/nhst/
- See also: Back safety - statpearls - NCBI bookshelf. — https://www.ncbi.nlm.nih.gov/books/NBK519066/
- See also: Emmi Educational Videos. Yale Health. — https://yalehealth.yale.edu/emmi-educational-videos